CLINICAL TRIAL: NCT06959706
Title: Phase 1, First-in-Human, Open-Label Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of TGW101 in Patients With Advanced Solid Tumors
Brief Title: Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of TGW101 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tagworks Pharmaceuticals BV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TGW101-101
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors
Keywords: Antibody-drug conjugates; Carcinoma; TGW101; TGW101-ADC; TRG001; TAG-72; Cancer
MeSH Terms: conditions — Carcinoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TGW101: Dose Escalation Cohorts (Experimental): Escalating doses of TGW101-anti-drug conjugate (ADC) will be administered via intravenous (IV) infusion followed by administration of TRG001. The treatment period continues until a reason for permanent discontinuation of treatment occurs.
  Interventions: Drug: TGW101
- TGW101: Enrichment Cohorts (Experimental): During Dose Escalation, additional participants may be enrolled to permit further evaluation of TGW101 to support selection of the optimal recommended dosing regimen(s) for expansion (RDE[s]). At the discretion of the Safety Oversight Committee (SOC), enrollment in enrichment cohorts may be limited to specific tumor type(s) based on assessment of clinical activity by the Sponsor in the dose escalation portion, and other nonclinical, translational, and clinical data.
  Interventions: Drug: TGW101

INTERVENTIONS:
Drug: TGW101 — TGW101 is a combination product comprising a chemically cleavable diabody drug conjugate (TGW101-ADC) and a corresponding small molecule chemical trigger (TRG001) administered separately.

SUMMARY:
The primary objectives of this study are to evaluate the safety and tolerability of TGW101 and determine the recommended dosing regimen(s) for further study. The secondary objectives are to assess pharmacokinetics and preliminary antitumor activity.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to any study procedures.
2. Males or females 18 years or older.
3. Histologically or cytologically confirmed diagnosis of a solid tumor malignancy listed below, with radiographic evidence of disease progression based on Response Evaluation Criteria in Solid Tumors (RECIST v1.1), or for castration resistant prostate cancer (CRPC), Prostate Cancer Clinical Trials Working Group 3, after most recent treatment and locally advanced or metastatic disease at Screening:

   1. Breast cancer (all subtypes).
   2. Castrate-resistant prostate cancer.
   3. Cervical cancer.
   4. Endometrial cancer.
   5. Esophageal, adenocarcinoma only.
   6. Gastric/gastroesophageal junction (GEJ).
   7. Non-squamous cell carcinoma of the head and neck, e.g., salivary gland neoplasms, with the exception of adenoid cystic carcinoma.
   8. Non-small cell lung cancer, adenocarcinoma only.
   9. Ovarian.
4. Refractory disease, intolerance to, or documented refusal of available standard therapy(ies) known to provide clinical benefit for the participant's solid tumor malignancy per Investigator judgment.
5. At least 1 measurable lesion per RECIST v1.1 except for participants with bone-only metastatic disease.
6. Biopsy pretreatment; if not possible, archival tissue block (preferred) or unstained formalin-fixed paraffin-embedded slides required.
7. Eastern Cooperative Oncology Group Performance Status 0-1.
8. Life expectancy of > 3 months in the opinion of the Investigator.
9. Adequate hepatic, hematologic, and renal function.

Exclusion Criteria:

1. Active second malignancy or history of another malignancy within the last 2 years, with the exception of: treated non-melanoma skin cancers; treated carcinoma in situ (e.g., breast and cervix); controlled superficial carcinoma of the urinary bladder; T1a or b carcinoma of the prostate; papillary thyroid carcinoma Stage I treated surgically for cure.
2. Known symptomatic brain metastases.
3. Significant cardiovascular disease within 6 months prior to starting study drug.
4. Evidence of an active systemic bacterial, fungal, or viral infection requiring treatment.
5. Grade ≥ 2 peripheral neuropathy.
6. Major surgery within 4 weeks prior to starting study drug.
7. Prior solid organ or bone marrow progenitor cell transplantation.
8. Prior high-dose chemotherapy requiring stem cell rescue.
9. Anticancer therapy within 28 days or within 5 half-lives (whichever is shorter) prior to starting study drug.
10. Palliative radiation therapy within 14 days prior to starting study drug.
11. Live vaccine within 28 days prior to starting study drug.
12. Pregnant or a breastfeeding postpartum female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events (AEs) | Up to approximately 10 months
Number of Participants Experiencing Dose-limiting Toxicities (DLTs) | Up to Day 21
Number of Participants Experiencing Cycle Delay | Up to approximately 10 months
Number of Participants Experiencing Dose Reduction | Up to approximately 10 months
RDE of TGW101 | Up to approximately 10 months

SECONDARY OUTCOMES:
Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast) of TGW101-ADC and TRG001 | Up to approximately 10 months
Area Under the Concentration-time Curve From Time Zero to the end of the Dosing Interval (AUCtau) of TGW101-ADC and TRG001 | Up to approximately 10 months
Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf) of TGW101-ADC and TRG001 | Up to approximately 10 months
Maximum Concentration (Cmax) of TGW101-ADC and TRG001 | Up to approximately 10 months
Trough Concentration (Ctrough) of TGW101-ADC and TRG001 | Up to approximately 10 months
Time to Maximum Concentration (Tmax) of TGW101-ADC and TRG001 | Up to approximately 10 months
Apparent Terminal Elimination Half-life (t1/2) of TGW101-ADC and TRG001 | Up to approximately 10 months
Steady-state Volume of Distribution (Vss) of TGW101-ADC and TRG001 | Up to approximately 10 months
Clearance (CL) of TGW101-ADC and TRG001 | Up to approximately 10 months
Accumulation Index of TGW101-ADC and TRG001 | Up to approximately 10 months
Overall Response Rate (ORR) | Up to approximately 10 months
Duration of Response (DOR) | Up to approximately 10 months
Progression-free Survival (PFS) | Up to approximately 10 months
Overall Survival (OS) | Up to approximately 10 months
Number of Participants Experiencing Antidrug Antibodies (ADAs) Against TGW101-ADC | Up to approximately 10 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Honor Health, Scottsdale, Arizona
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Dallas, Irving, Texas
  - NEXT San Antonio, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No